CLINICAL TRIAL: NCT01628926
Title: A Double-Blind, 3-Arm, Parallel Group, Placebo- and Ropinirole-Controlled Study for SPM 962 in Advanced Parkinson's Disease Patients With Concomitant Treatment of L-dopa
Brief Title: A Placebo- and Ropinirole-Controlled Study for SPM 962 in Advanced Parkinson's Disease Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 243-08-001; JapicCTI-090888 (Other: JAPIC)
Record Dates: First submitted 2012-06-24; First posted 2012-06-27 (Estimated); Results first posted 2014-05-23 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-04

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — ropinirole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- SPM 962 (Experimental): SPM 962 transdermal patch
  Interventions: Drug: SPM 962
- Ropinirole (Active Comparator): Ropinirole tablet
  Interventions: Drug: Ropinirole
- Placebo (Placebo Comparator): SPM962 placebo patch and Ropinirole placebo tab
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPM 962 — SPM 962 transdermal patch once a daily up to 36.0 mg/day
  Arms: SPM 962
Drug: Ropinirole — Ropinirole oral administration TID up to 15.0 mg/day
  Arms: Ropinirole
Drug: Placebo — SPM962-placebo patch and Ropinirole-placebo tab
  Arms: Placebo

SUMMARY:
* To demonstrate the non-inferiority of SPM 962 to ropinirole in terms of efficacy in order to confirm clinical value of SPM 962.
* To demonstrate the superiority of SPM 962 to placebo in terms of efficacy.
* To investigate the tolerability and safety of SPM 962 up to 36.0 mg/day.

ELIGIBILITY:
Inclusion Criteria:

* Subject diagnosed as having Parkinson's disease in accordance with "Diagnostic Criteria established by the Research Committee of MHLW-specified Intractable Neurodegenerative Diseases (1995)".
* Subject is 30 and more and less than 80 years of age at the time of informed consent.
* Hoehn & Yahr stage 2-4 (on time).
* Total UPDRS Part 3 score is over 10 at screening test (on time).
* Subject is on a stable dose of L-dopa with no change in daily dose or dosing regimen for at least 28 days prior to the initial treatment of SPM 962.
* Subject has any of the following problematic symptoms; 1) Wearing off phenomenon (including frozen gait at off time and dystonia at off time) 2) On and off phenomenon 3) Delayed-on and/or No-on phenomenon 4) Dyskinesia 5) Not well controlled with L-dopa.

Exclusion Criteria:

* Subject who has previously participated in a clinical trial of SPM962 and taken the investigational product (IP).
* Subject has psychiatric symptoms, e.g. confusion, hallucination, delusion, excitation, delirium, abnormal behavior at screening test or baseline.
* Subject whose SBP declines by at least 30 mmHg from supine to standing position based on the orthostatic hypotension assessment, or subject who develops orthostatic hypotension at baseline.
* Subject has a history of epilepsy, convulsion and other.
* Subject who has complications or a history of serious cardiac diseases or arrhythmia (eg, congestive heart failure of class 3 or 4 in the NYHA classification, second or third degree atrioventricular block, complete left bundle branch block, sick sinus syndrome, ventricular fibrillation, myocardial infarction within 12 months prior to the screening test, or a complication of angina pectoris).
* Subjects has QTc-interval >450 msec twice at screening. Subject has a the average QTc-interval from two ECGs >450 msec in males and >470 msec in females at baseline.
* Subject has congenital long QT syndrome.
* Subject whose serum potassium level is < 3.5mEq/L at the screening test.
* Subject has a total bilirubin >= 3.0 mg/dL or AST(GOT) or ALT(GPT) greater than 2.5 times of the upper limit of the reference range (or >= 100 IU/L) at screening test, or suffers complications of active phase of chronic hepatitis or liver cirrhosis.
* Subject has BUN >= 30 mg/dL or serum creatinine >= 2.0 mg/dl at screening test.
* Subject has a history of allergic reaction to topical agents such as transdermal patch.
* Subject has a history of known intolerance/hypersensitivity to ropinirole and/or adverse drug reactions that prevent subject from receiving treatment.
* Subject is pregnant or nursing or woman who plans pregnancy during the trial.
* Subject is receiving therapy with prohibited drug specified in the study protocol.
* Subject has a history of pallidotomy, thalamotomy, deep brain stimulation or fetal tissue transplant.
* Subject has dementia, including DLB and PDD (MMSE score <= 24 at screening).
* Subject who has a complication or history of malignant neoplastic disease, or received treatment for the disease within 12 months prior to the screening test.
* Subject is unable to give consent.
* Subject who is unable to properly record information in a diary.
* Subject is participating in another trial of IPs or received other IPs within 12 weeks prior to commencement of study treatment.
* Investigator judges that subject is inappropriate as a study subject with other reasons.

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2009-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyoji Imaoka, Mr, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (8):
- Japan (8):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Shikoku Region
  - Tohoku Region

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SPM 962 | Ropinirole | Placebo
Started | 168 | 167 | 85
Completed | 142 | 144 | 68
Not Completed | 26 | 23 | 17
Not completed — Adverse Event | 13 | 11 | 9
Not completed — Lack of Efficacy | 2 | 1 | 5
Not completed — Withdrawal by Subject | 6 | 4 | 2
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Discontinuation criteria | 3 | 4 | 0
Not completed — Physician Decision | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Population: 6 subjects were excluded. Met the exclusion criteria: 2 of SPM962, 1 of ropinirole Lack of efficacy observation: 2 of SPM962, 1 of Placebo
Groups:
- Total: Total of all reporting groups
Arm/Group | SPM 962 | Ropinirole | Placebo | Total
Number analyzed (Participants) | 164 | 166 | 84 | 414
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 71 | 52 | 28 | 151
  >=65 years | 93 | 114 | 56 | 263
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (8.8) | 67.0 (7.9) | 65.3 (7.9) | 65.8 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 98 | 42 | 243
  Male | 61 | 68 | 42 | 171
Region of Enrollment [Number; unit: participants]
  Japan | 164 | 166 | 84 | 414

OUTCOME MEASURES:

1. Primary Outcome: Unified Parkinson's Disease Rating Score (UPDRS) Part 3 Sum Score
Description: Mean change (LOCF) from baseline in UPDRS Part 3 sum score (on state) at 16 weeks after dosing.
  UPDRS is a scale for monitoring Parkinson's Disease-related disability and impairment. The UPDRS consists of the following four sub-scales. Part 1: Mentation, Part 2: Activities of Daily Living, Part 3: Motor, Part 4: Complications. Part 3 assesses 14 items. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: baseline, 16 weeks after dosing
Population: Full analysis set (FAS), last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM 962 | Ropinirole | Placebo
Number analyzed (Participants) | 164 | 166 | 84
Scores on a scale | -10.9 (8.1) | -9.5 (8.7) | -4.5 (9.7)

2. Secondary Outcome: UPDRS Part 3 Sum Score
Description: Mean change (LOCF) from baseline in UPDRS Part 3 sum score (on state) at 8 and 10 weeks after dosing.
  UPDRS Part 3 assesses 14 items. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: baseline, 8 and 10 weeks after dosing
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM 962 | Ropinirole | Placebo
Number analyzed (Participants) | 164 | 166 | 84
Scores on a scale
  8 weeks after dosing | -9.7 (7.2) | -8.4 (8.1) | -5.5 (8.3)
  10 weeks after dosing | -9.9 (7.1) | -8.8 (8.3) | -5.3 (9.0)

3. Secondary Outcome: UPDRS Part 2 Sum Score
Description: Mean change (LOCF) from baseline in UPDRS Part 2 sum score (average scores of on state and off state) at 16 weeks after dosing.
  UPDRS 2 assesses 13 items. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: Baseline, 16 weeks after dosing
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM 962 | Ropinirole | Placebo
Number analyzed (Participants) | 163 | 166 | 84
Scores on a scale | -3.6 (4.1) | -2.9 (3.5) | -1.3 (3.4)

4. Secondary Outcome: Off Time
Description: Mean change (LOCF) from baseline in off time at 16 weeks after dosing. Off-time is a state where L-Dopa becomes ineffective. Off-time was measured by patient diary in hours/day.
Time Frame: Baseline, 16 weeks after dosing
Population: FAS subjects with measurable off time data at baseline, LOCF
Measure: Mean (Standard Deviation); unit: Hours/day
Arm/Group | SPM 962 | Ropinirole | Placebo
Number analyzed (Participants) | 111 | 113 | 57
Hours/day | -1.3 (2.9) | -2.0 (3.0) | -0.4 (2.7)

5. Secondary Outcome: Parkinson's Disease Sleep Scale-2 (PDSS-2)
Description: Mean change (LOCF) from baseline in PDSS-2 sum score at 16 weeks after dosing. PDSS-2 is a scale for assessing sleep disorders in Parkinson's disease. PDSS consists of 15 questions about sleep and nocturnal disturbances. The score of each question ranges from 0 (never) to 4 (very frequent). The sum of each question serves as the scale score. Thus a decrease in the scores means improvement.
Time Frame: Baseline, 16 weeks after dosing
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM 962 | Ropinirole | Placebo
Number analyzed (Participants) | 162 | 165 | 81
Scores on a scale | -3.1 (6.8) | -3.4 (7.6) | -1.8 (7.0)

6. Secondary Outcome: On Time
Description: Mean change (LOCF) from baseline in on time at 16 weeks after dosing. On-time is a state where L-Dopa is effective. On-time was measured by patient diary in hours/day.
Time Frame: Baseline, 16 weeks after dosing
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Hours/day
Arm/Group | SPM 962 | Ropinirole | Placebo
Number analyzed (Participants) | 164 | 165 | 83
Hours/day | 1.3 (2.7) | 1.7 (2.9) | 0.2 (2.6)

7. Secondary Outcome: On Time Without Dyskinesia Disturbing Daily Activities
Description: Mean change (LOCF) from baseline in on time without dyskinesia disturbing daily activities at 16 weeks after dosing.
  On-time is a state where L-Dopa is effective. On-time was measured by patient diary in hours/day.
Time Frame: Baseline, 16 weeks after dosing
Population: FAS, LOCF Evaluation for this outcome measure was not possible, because only 22.6% (37/164), 12.7% (21/165), and 6.0% (5/83) of the subjects in the SPM 962, Ropinirole, and Placebo groups, respectively, had dyskinesia disturbing daily activities on either day from baseline until the end of titration/maintenance.
Measure: Mean (Standard Deviation); unit: Hours/day
Arm/Group | SPM 962 | Ropinirole | Placebo
Number analyzed (Participants) | 164 | 165 | 83
Hours/day | 1.1 (2.9) | 1.6 (3.0) | 0.3 (2.6)

8. Secondary Outcome: On Time With Dyskinesia Disturbing Daily Activities
Description: Mean change (LOCF) from baseline in on time with dyskinesia disturbing daily activities at 16 weeks after dosing (rate against on time).
Time Frame: Baseline, 16 weeks after dosing
Population: FAS, LOCF Evaluation for this outcome measure was not possible, because only 22.6% (37/164), 12.7% (21/165), and 6.0% (5/83) of the subjects in the SPM 962, Ropinirole, and Placebo groups, respectively, had dyskinesia disturbing daily activities on either day from baseline until the end of titration/maintenance period.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | SPM 962 | Ropinirole | Placebo
Number analyzed (Participants) | 37 | 21 | 5
Hours | 1.3 (11.0) | 0.6 (7.8) | -0.2 (1.4)

9. Secondary Outcome: Effective Rate in UPDRS Part 3 Sum Score
Description: Effective rate (percentage of subjects with 20% or 30% decrease) (LOCF) in UPDRS Part 3 sum score (on state) at 16 weeks after dosing.
Time Frame: Baseline, 16 weeks after dosing
Population: FAS, LOCF
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SPM 962 | Ropinirole | Placebo
Number analyzed (Participants) | 164 | 166 | 84
Percentage of participants
  ≥20% decrease | 80.5 [74.4 to 86.6] | 69.1 [62.0 to 76.1] | 56.6 [46.0 to 67.3]
  ≥30% decrease | 69.5 [62.5 to 76.6] | 60.6 [53.2 to 68.1] | 39.8 [29.2 to 50.3]

10. Secondary Outcome: Effective Rate in UPDRS Part 2 Sum Score
Description: Effective rate (percentage of subjects with 20% or 30% decrease) (LOCF) in UPDRS Part 2 sum score (average scores of on state and off state) at 16 weeks after dosing.
Time Frame: Baseline, 16 weeks after dosing
Population: FAS, LOCF
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SPM 962 | Ropinirole | Placebo
Number analyzed (Participants) | 163 | 166 | 84
Percentage of participants
  ≥20% decrease | 65.2 [57.9 to 72.6] | 56.7 [49.1 to 64.3] | 47.0 [36.3 to 57.7]
  ≥30% decrease | 55.9 [48.2 to 63.6] | 43.3 [35.7 to 50.9] | 28.9 [19.2 to 38.7]

11. Secondary Outcome: Effective Rate in Off Time
Description: Effective rate (percentage of subjects with 20% or 30% decrease) (LOCF) in off time at 16 weeks after dosing.
  On-time is a state where L-Dopa is effective. On-time was measured by patient diary in hours/day.
Time Frame: Baseline, 16 weeks after dosing
Population: FAS subjects with measurable off time data at baseline, LOCF
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SPM 962 | Ropinirole | Placebo
Number analyzed (Participants) | 111 | 113 | 57
Percentage of participants
  ≥20% decrease | 61.8 [52.7 to 70.9] | 65.5 [56.7 to 74.3] | 47.4 [34.4 to 60.3]
  ≥30% decrease | 55.5 [46.2 to 64.7] | 61.9 [53.0 to 70.9] | 40.4 [27.6 to 53.1]

12. Secondary Outcome: Clinical Global Impression (CGI)
Description: Change (LOCF) from baseline in CGI score. CGI improvement is a clinician-reported scale for assessing how much the patient's illness has improved or worsened from baseline.
  The scale scoring criteria are 1: very much improved, 2: much improved, 3: minimally improved, 4: no change, 5: minimally worse, 6: much worse, 7: very much worse. A decrease in the scores means improvement.
Time Frame: Baseline, 16 weeks after dosing
Population: FAS, LOCF
Measure: Number; unit: Percentage of Participants
Arm/Group | SPM 962 | Ropinirole | Placebo
Number analyzed (Participants) | 163 | 165 | 81
Percentage of Participants
  Decreased | 50.3 | 49.1 | 30.9
  Decreased (by at least 2 points) | 8.0 | 8.5 | 3.7
  Increased | 3.1 | 4.2 | 4.9
  Increased (by at least 2 points) | 0 | 0 | 0

13. Secondary Outcome: Dystonia (at an Early Hour)
Description: Change (LOCF) from baseline in occurrence of Dystonia (at an early hour).
Time Frame: Baseline, 16 weeks after dosing
Population: FAS, LOCF Evaluation for this outcome measure was not possible, because 87.1% (142/163), 88.5% (146/165), and 91.4% (74/81) of the subjects in the SPM 962, Ropinirole, and Placebo groups, respectively, had no dystonia in the day time at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | SPM 962 | Ropinirole | Placebo
Number analyzed (Participants) | 163 | 165 | 81
Percentage of participants
  Decreased | 10.4 | 10.9 | 7.4
  Decreased (by at least 2 events) | 1.8 | 4.2 | 2.5
  Increased | 1.2 | 3.0 | 3.7
  Increased (by at least 2 events) | 0 | 0.6 | 0

14. Secondary Outcome: Dystonia (in the Daytime)
Description: Change (LOCF) from baseline in occurrence of Dystonia (in the daytime).
Time Frame: Baseline, 16 weeks after dosing
Population: Appropriate interpretation for this outcome measure was not possible, because 87.1% (142/163), 88.5% (146/165), and 91.4% (74/81) of the subjects in the SPM 962, Ropinirole, and Placebo groups, respectively, had no dystonia in the day time at baseline.
Measure: Number; unit: Percentage of Participants
Arm/Group | SPM 962 | Ropinirole | Placebo
Number analyzed (Participants) | 163 | 165 | 81
Percentage of Participants
  Decreased | 8.6 | 7.9 | 3.7
  Decreased (by at least 2 events) | 3.7 | 5.5 | 2.5
  Increased | 3.7 | 2.4 | 4.9
  Increased (by at least 2 events) | 1.8 | 0.6 | 1.2

ADVERSE EVENTS:
Time Frame: 21 weeks
Arm/Group | SPM 962 | Ropinirole | Placebo
Serious Adverse Events (participants affected / at risk) | 7/168 | 5/167 | 6/85
Other Adverse Events (participants affected / at risk) | 140/168 | 99/167 | 40/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPM 962 (N=168) | Ropinirole (N=167) | Placebo (N=85)
Angina Pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric Ulcer Bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Carcinoma Gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Posture Abnormal (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Disease Parkinson's (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Cerebral Artery Embolism (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Delusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Caruncle Urethral (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Embolism Pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPM 962 (N=168) | Ropinirole (N=167) | Placebo (N=85)
Nausea (Gastrointestinal disorders) | 25 (27) | 23 (26) | 7 (8)
Vomiting (Gastrointestinal disorders) | 11 (15) | 11 (13) | 2 (2)
Application Site Reaction (General disorders) | 91 (93) | 30 (33) | 10 (11)
Application Site Pruritus (General disorders) | 6 (7) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 2 (2) | 3 (3)
Nasopharyngitis (Infections and infestations) | 28 (38) | 24 (29) | 13 (17)
Cystitis (Infections and infestations) | 3 (3) | 3 (3) | 4 (5)
Contusion (Injury, poisoning and procedural complications) | 7 (7) | 2 (2) | 6 (8)
Blood Creatine Phosphokinase Increased (Investigations) | 5 (5) | 6 (6) | 1 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5) | 2 (2)
Dyskinesia (Nervous system disorders) | 27 (28) | 23 (23) | 1 (1)
Hallucination Visual (Psychiatric disorders) | 13 (14) | 10 (10) | 3 (3)
Somnolence (Psychiatric disorders) | 11 (11) | 9 (9) | 2 (2)
Hallucination (Psychiatric disorders) | 3 (3) | 6 (6) | 0 (0)
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 3 (4)
Orthostatic Hypotension (Vascular disorders) | 5 (5) | 7 (8) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No